CLINICAL TRIAL: NCT02140775
Title: Return to Work Randomized Controlled Trial: Counseling After Fatigue Treatment in HIV/AIDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Callen-Lorde Community Health Center (Other)
Responsible Party: Principal Investigator, Martin McElhiney, Assistant Professor of Clinical Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6911
Record Dates: First submitted 2014-04-18; First posted 2014-05-16 (Estimated); Results first posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: HIV Infection; Fatigue
Keywords: HIV; AIDS; Fatigue; armodafinil; Unemployment
MeSH Terms: conditions — HIV Infections; Fatigue; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral Activation Counseling (Experimental): Behavioral Activation counseling is a manualized intervention adapted from a behavioral activation treatment for depression (BAT-D) and provides a basic foundation for behavior change. The individual sessions last one hour and are scheduled every two weeks. The counseling offers a brief, structured approach to identifying and scheduling activities in life areas to reduce avoidant behavior and increase activity level with the goal of achieving employment or enroll in training.
  Interventions: Behavioral: Behavioral Activation Counseling
- Supportive Counseling (Active Comparator): Supportive Counseling sessions will follow the same schedule and the Behavioral Activation Counseling, meeting for one hour every two weeks. The content of the sessions will be guided by the participant. The counselor will provide an accepting environment for the participant to explore his/her feelings about these topics.
  Interventions: Behavioral: Behavioral Activation Counseling

INTERVENTIONS:
Behavioral: Behavioral Activation Counseling — Behavioral Activation counseling is a manualized intervention adapted from a behavioral activation treatment for depression (BAT-D) and provides a basic foundation for behavior change. The individual sessions last one hour and are scheduled every two weeks. The counseling offers a brief, structured approach to identifying and scheduling activities in life areas to reduce avoidant behavior and increase activity level with the goal of achieving employment or enroll in training.
  Other Names: Behavioral Activation Therapy

SUMMARY:
The current study is a randomized clinical trial comparing Behavioral Activation counseling with supportive counseling for HIV+ participants presenting with clinically significant fatigue whose energy has improved with armodafinil, who have the goal of returning to work or vocational training but have not done so on their own. A second cohort of HIV+ participants without significant fatigue at baseline, but who also have the goal of returning to work, will also be randomized to either Behavioral Activation counseling or supportive counseling. In both cohorts, the primary outcome is level of success regarding an employment related goal.

DETAILED DESCRIPTION:
Despite the effectiveness of antiretroviral treatment to maintain or restore stable health, substantial numbers of HIV+ patients remain out of the mainstream and do not work. One important barrier is fatigue, which is prevalent and often disabling. After months to years of inertia and little activity, there is a need to rebuild one's life, which often requires support, guidance, time and reinforcement. Prior placebo controlled trials of modafinil and armodafinil to treat fatigue demonstrated efficacy. However, only 28% of those who wished to do so returned to work. Therefore the study team developed a manualized brief behavioral intervention, Behavioral Activation for Energy and Productivity (BA-PEP), derived from the validated Behavioral Activation Treatment for Depression, to be used in conjunction with armodafinil, with the primary goal of returning to work or vocational training.

The current study is a medication/behavioral intervention randomized controlled trial to test the efficacy of armodafinil/BA-PEP vs. armodafinil/Supportive Counseling (SC) in increasing energy, activity level and employment goal attainment for people with HIV/AIDS whose presenting problem is clinically significant fatigue and unmet work goals. The study will enroll HIV+ patients with clinically significant fatigue in a 4-week trial of armodafinil, those who experience improved energy will be eligible for the counseling program and randomized to BA-PEP or SC. To broaden the potential generalizability of the intervention, the study will also enroll HIV+ adults who do not meet criteria for clinically significant fatigue but who seek counseling to help them return to work. The study will be conducted at both New York State Psychiatric Institute and Callen Lorde Community Health Center, to examine intervention implementation within a real-world community clinic.

Primary aims: conduct a randomized clinical trial:

1. Determine if more participants in BA-PEP return to work compared to SC.
2. Determine if other outcome measures to assess behavioral activation and related dimensions, including the Environmental Reward Observation Scale [EROS], and Behavioral Activation for Depression Scale [BADS], differentiate response to BA-PEP and SC;
3. To identify predictors of success in work goal attainment, including moderator variables such as concurrent Axis I depression, age, education, health history and status, time since last employed full-time, and substance use history, as well as mediator variables (e.g. "dose" of counseling).

ELIGIBILITY:
Inclusion Criteria:

1. HIV+, age 18-70, and under the care of a medical provider
2. Clinically significant fatigue (Score of 4.5+ on Fatigue Severity Scale) and impairment on at least one category of role function (MOS) with duration of 3+ months (Does not apply to the cohort without fatigue)
3. Speaks English (reads English at high school level or shows comprehension in Evaluation to Consent procedure).
4. Able and willing to give informed consent
5. (Fecund Women): Uses barrier method of contraception
6. Patient seeks either work or job-related training

Exclusion Criteria:

1. Untreated Major Depression: (Structured Clinical Interview for Diagnostic and Statistical Manual IV (DSM-IV), (SCID) Depression Module;17-item Hamilton Rating Scale for Depression (HAM-D) >18).
2. Untreated hypogonadism, hypothyroidism or anemia (labs out of range).
3. Unstable medical condition
4. Left ventricular hypertrophy; symptomatic mitral valve prolapse (EKG; medical history)
5. Started testosterone in past 4 weeks
6. Started antidepressant medication in past 6 weeks
7. Substance abuse/dependence
8. Current clinically significant suicidal ideation
9. History or current psychosis or bipolar disorder
10. Pregnancy or breast feeding
11. Untreated insomnia (Score>3 on 3 HAM-D sleep items).
12. Currently taking stimulant medication of past non-responder to armodafinil

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2014-04-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith G Rabkin, Ph.D., MPH, Principal Investigator — Research Scientist VI
Locations (2):
- United States (2):
  - Callen-Lorde Community Health Center, New York, New York
  - New York State Psychiatric Institute, New York, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 138 patients who entered the study, 73 presented with significant fatigue and were started on armodafinil. Of those, 51 had an adequate response to the medication and were randomized to counseling. Another 65 patients did not have fatigue and were randomized directly to counseling. In total, 116 patients started counseling.
Groups:
- Behavioral Activation (BA) Counseling: Behavioral Activation counseling is a manualized intervention adapted from a behavioral activation treatment for depression (BAT-D) and provides a basic foundation for behavior change. The individual sessions last one hour and are scheduled every two weeks. The counseling offers a brief, structured approach to identifying and scheduling activities in life areas to reduce avoidant behavior and increase activity level with the goal of achieving employment or enroll in training.
- Supportive Counseling (SC): Supportive Counseling sessions will follow the same schedule and the Behavioral Activation Counseling, meeting for one hour every two weeks. The content of the sessions will be guided by the participant. The counselor will provide an accepting environment for the participant to explore his/her feelings about these topics.
Period: Overall Study
Arm/Group | Behavioral Activation (BA) Counseling | Supportive Counseling (SC)
Started | 87 | 29
Completed | 57 | 22
Not Completed | 30 | 7
Not completed — Withdrawal by Subject | 30 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Activation Counseling | Supportive Counseling | Total
Number analyzed (Participants) | 87 | 29 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (9.2) | 46 (10.0) | 47 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 87 | 29 | 116
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 9 | 24
  Not Hispanic or Latino | 72 | 20 | 92
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 11 | 35
  White | 62 | 18 | 80
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 29 | 116
Education [Mean (Standard Deviation); unit: years] | 14.8 (2.6) | 14.9 (2.2) | 14.8 (2.5)
Time since last worked regularly [Median (Inter-Quartile Range); unit: months] | 44 [3 to 300] | 36 [1 to 240] | 39 [1 to 300]
Receives Needs-based cash benefits [Count of Participants; unit: Participants] | 43 | 17 | 60
Has an AIDS diagnosis [Count of Participants; unit: Participants] | 44 | 15 | 59
Current Depression Diagnosis [Count of Participants; unit: Participants] | 38 | 6 | 44
Recent methamphetamine use problem [Count of Participants; unit: Participants] | 19 | 2 | 21

OUTCOME MEASURES:

1. Primary Outcome: Goal Attainment Scale - Modified (GAS): Responder (Score of 3 - Goal Achieved) vs. Non-Responder (Score of 1 or 2 - Goal NOT Achieved)
Description: Goal Attainment Scale - Prior to the beginning of counseling, the patient met with a member of the clinical team to develop an outcome GAS scale specific to their personal return to work goal. A goal was carefully established to be obtainable within the framework of 3-6 months, and to have observable anchors that could be scored on 3 outcome levels. A score of 3 indicates that they achieved their predetermined work goal and they were considered a "Responder" to the counseling. A score 2 indicates that some of the specific steps were taken towards the goal, but that it was not fully achieved. A score of 1 indicates that few or no steps were taken. Participants who scored 1 or 2 on their GAS scale were considered to be "Non-Responders."
  The Primary outcome presented below includes the number of participants who achieved their work-related goal (a score on the GAS scale of 3) and are considered RESPONDERS to counseling.
Time Frame: GAS Goal Responder vs. Goal Non-Responder will be assessed at Follow Up (3-6 months after the end of counseling)
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral Activation Counseling | Supportive Counseling
Number analyzed (Participants) | 57 | 22
Participants | 29 | 9
Statistical Analysis 1: Comparison: Behavioral Activation Counseling vs Supportive Counseling; A Chi-Square test was conducted between the treatment groups and the dichotomous outcome of successful achievement of employment goal; Test type: Superiority; p = .602, Chi-squared; degrees of freedom = 1

2. Secondary Outcome: Environmental Reward Observation Scale (EROS)
Description: This 10-item scale developed to assess changes in activity level and is based on the premise of response-contingent reinforcement.
  Score Range = 10 - 40 Higher scores suggest higher environmental reward.
Time Frame: EROS will be measured at Follow-up (3-6 months after the end of counseling)
Population: Not all participants completed the self-report measures at the Follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation Counseling | Supportive Counseling
Number analyzed (Participants) | 49 | 18
units on a scale | 27 (7) | 31 (8)
Statistical Analysis 1: Comparison: Behavioral Activation Counseling vs Supportive Counseling; Test type: Superiority; p = .066, t-test, 2 sided; Mean Difference (Final Values) = -3.74, 95% CI 2-sided [-7.75 to 0.26], Standard Error of Mean 2.00

3. Secondary Outcome: Behavioral Activation for Depression Scale (BADS)
Description: This 25 item scale total score is used to monitor change in Behavioral Activation (BA) protocols.
  Score Range = 0 - 150 Higher scores suggest greater activation and less avoidance, as well as less social and work impairment.
Time Frame: BADS will be measured Follow-up (3-6 months after the end of counseling)
Population: Not all participants completed the self-report measures at the Follow-up visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Activation (BA) Counseling | Supportive Counseling (SC)
Number analyzed (Participants) | 49 | 18
units on a scale | 99 (28) | 102 (27)
Statistical Analysis 1: Comparison: Behavioral Activation (BA) Counseling vs Supportive Counseling (SC); Test type: Superiority; p = .674, t-test, 2 sided; Mean Difference (Final Values) = -3.25, 95% CI 2-sided [-18.59 to 12.09], Standard Error of Mean 7.68

ADVERSE EVENTS:
Time Frame: The time frame included data collected from baseline until the final visit at follow up (3-6 months after the end of counseling)
Groups:
- Behavioral Activation Counseling: Behavioral Activation counseling is a manualized intervention adapted from a behavioral activation treatment for depression (BAT-D) and provides a basic foundation for behavior change. The counseling offers a brief, structured approach to identifying and scheduling activities in life areas to reduce avoidant behavior and increase activity level with the goal of achieving employment.
Arm/Group | Behavioral Activation Counseling | Supportive Counseling
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/29
Other Adverse Events (participants affected / at risk) | 0/87 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT02140775/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2013-07-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT02140775/SAP_001.pdf